CLINICAL TRIAL: NCT07186621
Title: Adjuvant Radiotherapy Combined With Sintilimab Versus Transarterial Chemoembolization (TACE) for Hepatocellular Carcinoma With Narrow Margins and High-Risk Features Following Resection: A Multi-center Phase III Randomized Controlled Trial
Brief Title: Adjuvant Radiotherapy of Sintilimab Versus TACE for HCC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Peking University People's Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Beijing 302 Hospital (Other); Beijing Ditan Hospital (Other); Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC5448
Record Dates: First submitted 2025-09-16; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma (HCC); Radiotherapy, Adjuvant; Immune Checkpoint Inhibitor; TACE; Narrow Margin
Keywords: hepatocellular carcinoma; radiotherapy; narrow margin; sintilimab; TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): The control group will receive the first TACE procedure within 4 months postoperatively, with the decision on administering a second TACE to be determined by the investigator based on the patient's condition and first TACE response assessment.
  Interventions: Procedure: TACE
- experiment group (Experimental): The experimental group will initiate radiotherapy within 4 months postoperatively with prescribed doses of 44-50Gy in 22-25 fractions to the tumor bed and 56-60Gy in 22-25 fractions to narrow-margin areas adjacent to major blood vessels, along with concurrent sintilimab 200mg q3w for 2 cycles followed by maintenance sintilimab 200mg q3w for 15 cycles (approximately 1 year total treatment duration) until disease progression or unacceptable toxicity.
  Interventions: Drug: Sintilimab; Radiation: radiotherapy

INTERVENTIONS:
Drug: Sintilimab — concurrent sintilimab 200mg q3w for 2 cycles followed by maintenance sintilimab 200mg q3w for 15 cycles (approximately 1 year total treatment duration) until disease progression or unacceptable toxicity
  Arms: experiment group
Radiation: radiotherapy — The experimental group will initiate radiotherapy within 4 months postoperatively with prescribed doses of 44-50Gy in 22-25 fractions to the tumor bed and 56-60Gy in 22-25 fractions to narrow-margin areas adjacent to major blood vessels
  Arms: experiment group
Procedure: TACE — The control group will receive the first TACE procedure within 4 months postoperatively, with the decision on administering a second TACE to be determined by the investigator based on the patient's condition and first TACE response assessment.
  Arms: control group

SUMMARY:
This study is an open-label, randomized controlled, multicenter, phase III clinical trial

DETAILED DESCRIPTION:
This study is an open-label, randomized controlled, multicenter, phase III clinical trial where participants are randomized in a 1:1 ratio to either the experimental or control group. The experimental group will initiate radiotherapy within 4 months postoperatively with prescribed doses of 44-50Gy in 22-25 fractions to the tumor bed and 56-60Gy in 22-25 fractions to narrow-margin areas adjacent to major blood vessels, along with concurrent sintilimab 200mg q3w for 2 cycles followed by maintenance sintilimab 200mg q3w for 15 cycles (approximately 1 year total treatment duration) until disease progression or unacceptable toxicity. The control group will receive the first TACE procedure within 4 months postoperatively, with the decision on administering a second TACE to be determined by the investigator based on the patient's condition and first TACE response assessment. The primary endpoint is 2-year recurrence-free survival (RFS) rate, while secondary endpoints include 2-year overall survival (OS) rate and incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. R0 resection of hepatocellular carcinoma (HCC) with a surgical margin <1 cm (determined by postoperative pathology, surgical records, and imaging).
2. Within 4 months after curative resection.
3. High-Risk Recurrence Factors (at least one required in addition to narrow margin): (1) Microvascular invasion (MVI) positive, tumor thrombus, or satellite nodules (2) Preoperative AFP >400 ng/mL (3) Tumor >5 cm with incomplete capsule
4. ≥18 and ≤80 years old.
5. ECOG score 0-1.
6. Child-Pugh Class: A5, A6, or B7.
7. Postoperative Contrast-enhanced MRI of the liver must be performed to exclude intrahepatic residual lesions.
8. HBV DNA and HCV RNA status do not affect eligibility, but if HBV DNA positive and/or HCV RNA positive: ALT must be <1.5× upper limit of normal (ULN). Antiviral therapy must be initiated.
9. Liver Function Tests (LFTs): ALT ≤2.5× ULN (if HBV/HCV positive, ALT ≤1.5× ULN). If ALT ≤1.5× ULN, AST ≤6× ULN (excluding AST elevation due to myocardial infarction). If ALT 1.5-2.5× ULN, AST ≤2.5× ULN.
10. No significant ECG abnormalities and no severe cardiac dysfunction.
11. Serum creatinine (CRE) and BUN ≤2.5× ULN.
12. Hb≥80g/L，ANC≥1.0×109 /L，PLT≥40×109 /L.
13. Written informed consent obtained.

Exclusion Criteria:

1. Vp3 or Vp4 portal vein tumor thrombus (PVTT) or Vv2/Vv3 inferior vena cava (IVC) tumor thrombus on preoperative imaging.
2. Previous anti-HCC therapies, including but not limited to: targeted therapy (e.g., tyrosine kinase inhibitors), immune checkpoint inhibitors (e.g., PD-1/PD-L1 inhibitors) or systemic chemotherapy
3. Distant metastasis before randomization.
4. Moderate to severe ascites unresponsive to medical management.
5. History of other malignancies, except: carcinoma in situ，early-stage papillary thyroid cancer or basal cell carcinoma of the skin
6. Previous radiotherapy involving the abdomen.
7. Significant cardiac, renal, or other major organ dysfunction.
8. Active Autoimmune Disease or Psychiatric Disorders.
9. HIV Infection.
10. Pregnant or breastfeeding women.
11. Currently enrolled in another interventional clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2027-07-09 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
2-year RFS | 2-year after randomization
  the percentage of patients who remain free of detectable cancer recurrence (local, regional, or distant) and alive for at least 2 years after randomization

SECONDARY OUTCOMES:
2-year OS | 2-year after randomization
  the percentage of patients who are still alive (from any cause) at 2 years after randomization
adverse events | up to 2 years after randomization
  any symptoms, signs, and laboratory examinations abnormality during the clinical trial

CONTACTS AND LOCATIONS:
Overall Officials: Shuhang Wang, Study Director — NCC, CICAMS
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No